CLINICAL TRIAL: NCT00409357
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose Ranging Study of SL77.0499-10 Once Daily Tablets in Patients With Lower Urinary Tract Symptoms Related to Benign Prostatic Hyperplasia (BPH)
Brief Title: Dose Ranging Study of Alfuzosin in Patients With Lower Urinary Tract Symptoms Related to Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5234
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: urinary tract
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SL77.0499-10 (alfuzosin hydrochloride)

SUMMARY:
The primary objective is to assess the dose-response relationship of SL77.0499 10 (alfuzosin hydrochloride) 5 mg, 10 mg, 15 mg, and placebo once daily during a 12-week oral administration period for the efficacy in patients with lower urinary tract symptoms (LUTS) related to BPH.

Secondary objectives are to assess the efficacy of each dose of alfuzosin as compared with placebo and to assess the safety of each dose of alfuzosin.

ELIGIBILITY:
Inclusion Criteria:

* suffering from LUTS related to BPH for at least 6 months;
* having an IPSS >13;
* having a urinary peak flow rate 5.0 to 12.0 mL/s for a voided volume of at least 150 mL;
* having a residual urine volume < or = 200 mL.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2004-11; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy assessment is the change from baseline in International Prostate Symptom Score (IPSS) total score at the end-of-study (EOS) visit.

SECONDARY OUTCOMES:
Efficacy: changes from baseline in IPSS total score by visit;·IPSS irritative and obstructive subscores,·urinary peak flow rate and residual urine volume at EOS and by visit.
Safety: adverse events, vital signs, laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan